CLINICAL TRIAL: NCT07124676
Title: Prospective Observational Study Comparing Two Classifications of Second-degree Perineal Tears in Spontaneous Vaginal Births, to Evaluate Their Correlation With Postpartum Clinical Outcomes.
Brief Title: Prospective Study Comparing Two Classification Systems for Second-degree Vaginal Tears During Spontaneous Childbirth to Assess Their Ability to Predict Postpartum Complications.
Acronym: LAC-VAG-2025
Status: Not yet recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, Researcher, University of Campania Luigi Vanvitelli
Other Study IDs: 0016346/i
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Vaginal Laceration During Delivery
Keywords: vaginal laceration; delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with spontaneous second-degree perineal tears: Participants are women who have a spontaneous vaginal birth and sustain a spontaneous second-degree perineal tear. Each tear is classified according to both the Scandinavian (Macedo et al., 2022) and De Simone systems during routine postpartum examination. No experimental intervention is performed; outcomes are collected through clinical records, postpartum examination, ultrasound, and validated questionnaires (FSFI).

SUMMARY:
Second-degree perineal tears are one of the most common complications during vaginal childbirth. These injuries involve the muscles of the perineum but do not affect the anal sphincter. Although frequent, they vary greatly in severity, and their short- and long-term consequences can include pain, bleeding, hidden muscle damage, and sexual function problems.

Currently, there is no widely used, detailed system to sub-classify these tears, which makes it harder to study their relationship with postpartum complications and to guide follow-up care. Two classification systems have been proposed:

The Scandinavian classification (Macedo et al., 2022), which grades second-degree tears based on the percentage of the perineal body involved (2A: <50%, 2B: >50%, 2C: entire perineal body and/or large vaginal extension).

The De Simone classification, which describes tears according to their extension along the vaginal wall (lower third, middle third, upper third/fornices) and muscle involvement, with specific codes for isolated locations.

This prospective, single-center observational study at AOU Vanvitelli will enroll 482 women who have a spontaneous vaginal delivery and a spontaneous second-degree perineal tear. Each tear will be independently classified according to both systems, without any additional procedures beyond routine clinical care.

The primary aim is to determine which classification better correlates with important postpartum outcomes: significant drop in hemoglobin levels, moderate-to-severe perineal pain (VAS ≥5), occult lesions detected by postpartum perineal ultrasound, and abnormal Female Sexual Function Index (FSFI) scores at follow-up.

By directly comparing these two systems in the same population, the study seeks to identify whether a more detailed classification can improve prediction of complications, guide patient counseling, and inform postpartum follow-up. The findings may contribute to better standardization in describing these tears and improved care for women after childbirth.

DETAILED DESCRIPTION:
Second-degree perineal tears are among the most frequent complications of spontaneous vaginal delivery, involving the perineal muscles without damage to the anal sphincter complex. Despite their high incidence, these tears vary greatly in depth, length, and anatomical involvement, which may affect postpartum pelvic floor health, pain, bleeding, and sexual function. Current standard classification systems, such as that recommended by the Royal College of Obstetricians and Gynaecologists (RCOG), do not provide subcategories for second-degree tears, potentially limiting accurate prognostic assessment.

Two more detailed systems have been proposed:

Scandinavian classification (Macedo et al., 2022) - subdivides second-degree tears based on the percentage of the perineal body affected:

2A: <50% of the perineal body, with or without lower vaginal tear ≤2 cm.

2B: >50% of the perineal body, with or without lower vaginal tear ≤2 cm.

2C: entire perineal body, with or without lower vaginal tear >2 cm. Vaginal extensions >4 cm from the tear margin are also documented.

De Simone classification - describes second-degree tears according to their vaginal extension and muscle involvement:

2a: lower third of the vagina with muscle involvement (includes uncomplicated episiotomy).

2b: extension from the lower to the middle third of the vagina.

2bx: isolated tear of the middle third of the vagina.

2c: extension from the lower to the upper third (including fornices).

2cx: isolated tear of the upper third (including fornices).

Evidence comparing these systems in terms of clinical outcome prediction is lacking.

Study Design This is a prospective, single-center, observational cohort study conducted at AOU Vanvitelli - UOC di Ostetricia e Ginecologia. The study will enroll 482 women undergoing spontaneous vaginal delivery who sustain a spontaneous second-degree perineal tear.

No experimental intervention is performed; classification occurs during routine postpartum examination.

All eligible tears will be classified independently by two trained operators using both classification systems.

Data will be collected on hemoglobin change, perineal pain, postpartum ultrasound findings, and FSFI scores.

Objectives

Primary Objective: Compare the diagnostic accuracy of the Scandinavian vs. De Simone classification systems in predicting postpartum complications.

Secondary Objectives: Evaluate the association of each tear subtype with:

Postpartum hemoglobin reduction

Perineal pain (VAS ≥5)

Occult lesions detected by perineal ultrasound

Pathological FSFI scores

Population

Inclusion Criteria:

Spontaneous vaginal birth at AOU Vanvitelli

Spontaneous second-degree perineal tear

Signed informed consent

Exclusion Criteria:

Episiotomy or operative vaginal delivery

Obstetric conditions preventing spontaneous birth

Age <18 years

Sample Size and Statistical Plan Based on Italian national data (SIGO 2024) estimating a 35% incidence of second-degree tears and internal delivery room records showing 29% incidence, a sample size of 482 women provides 80% power at α = 0.05 to detect clinically meaningful differences in outcome prediction between classifications.

Analysis:

Descriptive statistics for baseline and outcome variables.

Tests for normality (Shapiro-Wilk) and graphical inspection.

Comparisons between subtypes:

t-test or ANOVA for normally distributed continuous variables (Bonferroni/Tukey post-hoc).

Mann-Whitney U or Kruskal-Wallis for non-normal data.

Chi-square or Fisher's exact test for categorical variables.

Multivariate logistic regression to identify independent predictors of complications, adjusting for age, parity, neonatal weight, and labor duration. Multicollinearity will be assessed via VIF; model fit via Hosmer-Lemeshow; discrimination via AUC.

Data Quality and Management

Data will be entered into a secure electronic database with predefined value ranges and logical consistency checks.

Source data verification will be performed by cross-checking electronic records with delivery notes and patient charts.

Missing data will be flagged; analyses will specify handling strategies (complete case vs. multiple imputation depending on pattern/extent).

Variables are coded in a standardized data dictionary; clinical classifications follow published definitions (Macedo et al., 2022; De Simone).

All study personnel will follow SOPs for recruitment, consent, classification, data collection, entry, and storage.

Ethics and Safety The study is non-interventional and poses no additional risk beyond routine postpartum care. All procedures comply with the Declaration of Helsinki (2008) and Good Clinical Practice (GCP). Participants incur no costs and receive no financial incentives.

ELIGIBILITY:
Inclusion Criteria:

Female at birth.

Age 18 years or older.

Spontaneous vaginal delivery

Presence of a spontaneous second-degree perineal tear, confirmed on postpartum examination.

Able and willing to provide informed consent to participate in the study.

Exclusion Criteria:

Delivery involving episiotomy.

Operative vaginal delivery (forceps or vacuum).

Obstetric or medical conditions preventing spontaneous vaginal delivery.

Inability to understand study procedures or complete follow-up assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals identifying as female at birth are eligible to participate, as the study population consists of women experiencing spontaneous vaginal delivery with spontaneous second-degree perineal tears.
Study Population: Women giving birth, who experience a spontaneous vaginal delivery resulting in a spontaneous second-degree perineal tear. Participants are recruited consecutively from the hospital's maternity ward during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
hemoglobin reduction | within 48 hours postpartum
  significant hemoglobin reduction (>2 g/dL from pre- to post-delivery)
moderate-to-severe perineal pain | within 48 hours postpartum
  VAS ≥ 5
pathological Female Sexual Function Index (FSFI) total score | within 48 hours after the delivery
  FSFI total score modification after vaginal laceration.

SECONDARY OUTCOMES:
occult perineal or vaginal muscle lesions | within 7 days postpartum for ultrasound assessment; at 3 months postpartum for FSFI evaluation.
  occult perineal or vaginal muscle lesions on postpartum perineal ultrasound;

CONTACTS AND LOCATIONS:
Locations (1):
- Universita degli studi della Campania "Luigi Vanvitelli" - dipartimento della donna, bambino e chirurgia generale e specialistica,, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policies and ethical considerations regarding the protection of participants' privacy.

REFERENCES:
- [Background] Kryter KD. Evaluation of hearing handicap. The American Academy of Otolaryngology and American Council of Otolaryngology (AA0-ACO). J Am Acad Audiol. 1998 Apr;9(2):141-6. PMID 9564677